CLINICAL TRIAL: NCT04134117
Title: Pilot Study of Tisagenlecleucel, CD19-targeted Chimeric Antigen Receptor (CAR) T Cells, in Patients With Primary Central Nervous System Lymphoma
Brief Title: Tisagenlecleucel In Primary CNS Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Matthew J. Frigault, M.D. (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Matthew J. Frigault, M.D., Sponsor Investigator, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-319
Record Dates: First submitted 2019-10-18; First posted 2019-10-22 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Primary CNS Lymphoma; Refractory Primary CNS Lymphoma; Relapsed Primary CNS Lymphoma
Keywords: Primary CNS Lymphoma; Refractory Primary CNS Lymphoma; Relapsed Primary CNS Lymphoma
MeSH Terms: interventions — tisagenlecleucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tisagenlecleucel (Experimental): Study procedures include screening for eligibility and study treatment including, leukapheresis, evaluations, and follow up visits.
  - Tisagenlecleucel will be administered intravenously as a one-time rapid infusion predetermined dose following lymphodepleting chemotherapy.
  Interventions: Biological: Tisagenlecleucel

INTERVENTIONS:
Biological: Tisagenlecleucel — One time single predetermined dose level CAR-positive T cells will be utilized based on the FDA approved product label.
  Other Names: KYMRIAH

SUMMARY:
In this study, is researching the safety of tisagenlecleucel in participants with primary central nervous system lymphoma. .

-The name of the study intervention is tisagenlecleucel.

DETAILED DESCRIPTION:
This research study is a Pilot Study, which is the first time investigators are examining this intervention in people with primary central nervous system lymphoma.

* The name of the study intervention is tisagenlecleucel. Tisagenlecleucel is an investigational treatment that uses the participants own immune cells, called T cells, to try to kill the cancerous cells
* The research study procedures include screening for eligibility and study treatment including, leukapheresis, evaluations, and follow up visits.
* The study treatment will be one day and participants will be followed for up to 2 years.
* It is expected that about 12 people will take part in this research study

ELIGIBILITY:
Inclusion Criteria:

Primary CNS Lymphoma in high risk elderly patients

* New diagnosis of primary CNS lymphoma.
* Voluntarily sign informed consent form(s)
* ≥60 years of age at the time of signing informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2
* Have failed or are unable to tolerate definitive first-line methotrexate based therapy as defined by:

  * Grade 3+ AKI and/or transaminitis preventing repeat treatment exposure and/or,
  * Failure to achieve a complete response (per IPCG) following two cycles of first line therapy,

    --- Definitive first-line therapies must include high dose methotrexate-based therapy but may also include temozolomide, high dose cytarabine, pemetrexed, lenalidomide, ibrutinib and rituximab.
  * Whole-brain irradiation, lenalidomide monotherapy and ibrutinib monotherapy are considered first line therapy if patient was not eligible for methotrexate-based chemotherapy at time of initial treatment but now meets study eligibility criteria.
* Adequate absolute lymphocyte count (ALC > 500 cells/ul) within one week of apheresis.
* Adequate bone marrow function defined by absolute neutrophil count (ANC) >1000 cells/mm3without growth factor support, and untransfused platelet count >50,000 mm3 within 7 days.
* Left ventricular ejection fraction >40%
* Adequate hepatic function defined by aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) <2.5 × upper limit of normal (ULN) and direct bilirubin <1.5 × ULN
* Adequate renal function defined by creatinine clearance >30 ml/min using the Cockcroft-Gault formula
* International ratio (INR) or partial thromboplastin time (PTT) <1.5 × ULN, unless on a stable dose of anticoagulant for a thromboembolic event.
* The effects of tisagenlecleucel T cells on the developing human fetus are unknown. For this reason, women of child-bearing potential and men with partners of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to leukapheresis for at least 1-year post tisagenlecleucel infusion and until CAR T cells are no longer present by qPCR on two consecutive tests. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men with partners of childbearing potential treated or enrolled on this protocol must also agree to use adequate contraception prior to leukapheresis and until 4 months after tisagenlecleucel T cells administration.
* Ability and willingness to adhere to the study visit schedule and all protocol requirements

Relapsed/Refractory Primary CNS Lymphoma

* Diagnosis of relapsed/refractory PCNSL having received at least one prior line of CNS directed therapy.
* Voluntarily sign informed consent form(s)
* ≥18 years of age at the time of signing informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Adequate absolute lymphocyte count (ALC > 500 cells/ul) within one week of apheresis.
* Adequate bone marrow function defined by absolute neutrophil count (ANC) >1000 cells/mm3without growth factor support, untransfused platelet count >50,000 mm3, and untransfused hemoglobin >9 g/dL.
* Left ventricular ejection fraction >40%
* Adequate hepatic function defined by aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) <2.5 × upper limit of normal (ULN) and direct bilirubin <1.5 × ULN
* Adequate renal function defined by creatinine clearance >30 ml/min using the Cockcroft-Gault formula
* International ratio (INR) or partial thromboplastin time (PTT) <1.5 × ULN, unless on a stable dose of anticoagulant for a thromboembolic event.
* The effects of tisagenlecleucel T cells on the developing human fetus are unknown. For this reason, women of child-bearing potential and men with partners of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to leukapheresis for at least 1-year post tisagenlecleucel infusion and until CAR T cells are no longer present by qPCR on two consecutive tests. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men with partners of childbearing potential treated or enrolled on this protocol must also agree to use adequate contraception prior to leukapheresis and until 4 months after tisagenlecleucel T cells administration.
* Ability and willingness to adhere to the study visit schedule and all protocol requirements

Inclusion Criteria for Lymphodepletion/Cell Infusion:

* No Active, uncontrolled, systemic bacterial, viral, or fungal infection.
* Adequate renal function defined by creatinine clearance >30 ml/min using the Cockcroft-Gault formula

Exclusion Criteria:

* Prior treatment with an any investigational cellular therapy.
* Ongoing treatment with chronic immunosuppressants (e.g., cyclosporine). Systemic steroids are allowed up to a dose of dexamethasone 4mg daily or equivalent.
* Ongoing systemic immunosuppression for acute and/or chronic GVH as a result of previous allogeneic bone marrow transplant.
* Significant co-morbid condition or disease which in the judgment of the Principal Investigator would place the subject at undue risk or interfere with the study; examples include, but are not limited to, cirrhotic liver disease, sepsis, and/or recent significant traumatic injury.
* Active, uncontrolled, systemic bacterial, viral, or fungal infection.
* Active hepatitis B or hepatitis C infection.
* HIV infection.
* Subjects with a history of class III or IV congestive heart failure or non- ischemic cardiomyopathy.
* Subjects with second malignancies if the second malignancy has required therapy in the last 3 years or is not in complete remission; exceptions to this criterion include successfully treated non-metastatic basal cell or squamous cell skin carcinoma, or prostate cancer that does not require therapy other than hormonal therapy.
* Pregnant or lactating women
* Live virus vaccines within 2 weeks prior to planned start of lymphodepleting chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-04-14 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE Criteriaand ASTCT 2018 (CRS/NT) | 12 Months

SECONDARY OUTCOMES:
Objective disease response to tisagenlecleucel | 1 Month
  IPCG response criteria.
Objective disease response to tisagenlecleucel | 3 Months
  IPCG response criteria.
Objective disease response to tisagenlecleucel | 6 months
  IPCG response criteria.
Objective disease response to tisagenlecleucel | 12 months
  IPCG response criteria.
Overall Survival Rate | 15 years
  Kaplan-Meier method
Progression Free Survival Rate | from the date of assignment until the date of first documented progression or date of deathfrom any cause, whichever comes first, assessed up to 100 months
  Kaplan-Meier method

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J. Frigault, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: MGH - Contact the Partners Innovations team at http://www.partners.org/innovation

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-08): https://cdn.clinicaltrials.gov/large-docs/17/NCT04134117/Prot_SAP_000.pdf